CLINICAL TRIAL: NCT00521963
Title: Interventional Study: Administration of Intraarticular Injection of Infliximab in Patients With Inflammatory Arthritis Who Failed Intraarticular Injection of Corticosteroids
Brief Title: Intraarticular Injection of Infliximab
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: poor accrual
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Bnai Zion Medical Center (Other Government); Carmel Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0088-07-EMC
Record Dates: First submitted 2007-08-17; First posted 2007-08-28 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Arthritis
Keywords: Intraarticular injection; Infliximab
MeSH Terms: conditions — Arthritis | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- E (Experimental)
  Interventions: Biological: Intraarticular injection of infliximab

INTERVENTIONS:
Biological: Intraarticular injection of infliximab — A single injection of 100 mg of infliximab
  Other Names: Remicade

SUMMARY:
Intra-articular (IA) injection of medication is a common procedure in the management of joint disorders. In particular, the procedure is effective in the treatment of inflammatory conditions, with long acting corticosteroids most commonly used. These agents have been shown to reduce the signs and symptoms of inflammation, expressed primarily in the synovium of the joint, and are probably capable of slowing the progression of damage to joint cartilage and bone in some of these inflammatory conditions. Arthritis that is refractory to IA corticosteroid injections may respond to surgical, chemical, or, radioisotope synovectomy, procedures in which the inflamed synovial tissue is eradicated. It has been noted that infliximab, a monoclonal antibody directed to Tumor Necrosis Factor (TNF) - α, has high affinity for the TNF-α rich inflamed synovium. Recently, clinical benefit from IA injections of infliximab has been reported in some cases that were refractory to IA injections of corticosteroids. Similarly, the effectiveness of IA infliximab in suppression of joint inflammation has also been demonstrated in patients who could not receive systemic therapy with infliximab. These reports examined the effect of a single injection of infliximab100 mg injected into a large inflamed joint or 2 IA injections 24 hours apart.

We propose to further evaluate the use of IA infliximab in patients with intractable knee monoarthritis, explore the optimal mode of its employment, and assess the degree of infliximab systemic absorption from the IA injection. In a pilot study 40 knees will be evaluated, 20 injected with infliximab and 20 injected with a corticosteroid comparator reflecting the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Have non-infectious monoarthritis of the knee and with inadequate response to IA injection of corticosteroids, at least 3 months before enrollment.

or

* Have oligo or polyarthritis controlled by disease modifying agents (DMARDs) but with residual 1-2 inflamed joints, one of which is a knee with inadequate response to IA injection of corticosteroids within 3 months
* Have negative PPD skin test.
* Have no evidence of TB on chest x-ray.
* Be negative for HBsAg and HCV.
* No evidence of infectious arthritis

Exclusion Criteria:

* Known allergy to infliximab.
* Known allergy to lidocaine.
* Pregnant.
* Female patients with childbearing potential who do not practice effective methods of contraception.
* Suffer from a chronic infection.
* On systemic anti TNF-α or other biologic agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
suppression of inflammation | 12 weeks

SECONDARY OUTCOMES:
Amount of systemic absorbtion | 2,4,8,12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Mader, MD, Principal Investigator — Ha'Emek Medical Center, Afula, Israel
Locations (2):
- Israel (2):
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center and Lin outpatient service, Haifa

REFERENCES:
- [Background] Schatteman L, Gyselbrecht L, De Clercq L, Mielants H. Treatment of refractory inflammatory monoarthritis in ankylosing spondylitis by intraarticular injection of infliximab. J Rheumatol. 2006 Jan;33(1):82-5. Epub 2005 Nov 15. PMID 16292792
- [Background] Conti F, Priori R, Chimenti MS, Coari G, Annovazzi A, Valesini G, Signore A. Successful treatment with intraarticular infliximab for resistant knee monarthritis in a patient with spondylarthropathy: a role for scintigraphy with 99mTc-infliximab. Arthritis Rheum. 2005 Apr;52(4):1224-6. doi: 10.1002/art.20979. PMID 15818709
- [Background] Nikas SN, Temekonidis TI, Zikou AK, Argyropoulou MI, Efremidis S, Drosos AA. Treatment of resistant rheumatoid arthritis by intra-articular infliximab injections: a pilot study. Ann Rheum Dis. 2004 Jan;63(1):102-3. doi: 10.1136/ard.2003.006981. No abstract available. PMID 14672902